CLINICAL TRIAL: NCT01184326
Title: An Expanded Phase I Study of Pazopanib and Everolimus in Patients With Advanced Solid Tumors and Previously Treated Advanced Urothelial Cancer
Brief Title: Expanded Phase I Pazopanib and Everolimus in Advanced Solid Tumors and Previously Treated Advanced Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Mark Pomerantz, MD, Assistant Professor of Medicine, Harvard Medical School, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-166
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor; Kidney Cancer
Keywords: RAD001; pazopanib; everolimus; advanced cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — pazopanib; Everolimus

STUDY DESIGN:
Intervention Model Description: This is a Phase I study with multiple arms related to planned dose escalation.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 0: Everolimus 5mg + Pazopanib 600 mg (Experimental): Everolimus 5mg + Pazopanib 600 mg once daily for 28 days each cycle Participants were treated until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: pazopanib; Drug: everolimus
- Dose Level -1: Everolimus 5mg + Pazopanib 400 mg (Experimental): Everolimus 5mg + Pazopanib 400 mg once daily for 28 days each cycle Participants were treated until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: pazopanib; Drug: everolimus
- All Phase I Dose Expansion Participants (Experimental): All phase I dose expansion participants received Everolimus 5mg and Pazopanib at the maximum tolerated dose established in the dose finding part of the study.
  Interventions: Drug: pazopanib; Drug: everolimus
- All Phase I Participants (Experimental): All phase I participants received Everolimus 5mg and Pazopanib according to the established dose escalation schedule or the maximum tolerated dose established in the dose finding part of the study.
  Interventions: Drug: pazopanib; Drug: everolimus

INTERVENTIONS:
Drug: pazopanib
  Other Names: Votrient
Drug: everolimus
  Other Names: RAD001

SUMMARY:
This research study is evaluating the combination of pazopanib and everolimus in patients that have a malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective, or metastatic or locally advanced unresectable kidney cancer. In this research study the investigators are testing the safety of the combination of pazopanib and everolimus and finding the appropriate doses to use for further studies.

DETAILED DESCRIPTION:
This protocol has two parts, Phase I Dose Finding and Phase 1 Expansion. Once the maximum tolerated dose has been identified in the Phase I Dose Finding portion, a Phase I expansion cohort of patients with metastatic or locally advanced unresectable kidney cancer will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Participants must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effected.
* Expansion Cohort Only: Participants must have histologically or cytologically confirmed metastatic or locally advanced unresectable kidney cancer.
* Expansion Cohort Only: Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension at 20mm or greater with conventional techniques or as 10mm or greater with spiral CT.
* Expansion Cohort Only: Previously treated with at least one anti-angiogenic agent, including but not limited to bevacizumab, sunitinib, or sorafenib. No more than 4 lines of prior systemic therapy for kidney cancer, mTOR pathway inhibitors other than RAD001 are allowed.
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG performance status of 0 or 1
* Normal organ and marrow function as outlined in the protocol
* Able to swallow oral medications
* Resolution of any pre-existing toxicity from prior therapy to NCI CTCAE v4.0 grade 1 or less
* Women are eligible to participate if she is of non-child bearing potential or agrees to use adequate contraception
* Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
* A male with a female partner of childbearing potential must use a barrier method of contraception or abstinence during the study

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or thos who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Current treatment with leuprolide or other GnRH agonists is permitted on the Phase 1 portion of the study.
* Participants may not be receiving any other study agents.
* Prior RAD001 or pazopanib therapy
* History of clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 weeks prior to the first dose of study drug.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or everolimus
* History of any of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting; myocardial infarction; unstable angina; coronary artery by-pass graft surgery; symptomatic peripheral vascular disease; Class III or IV congestive heart failure
* Poorly controlled hypertension
* History of cerebrovascular accident, pulmonary embolism, or untreated deep venous thrombosis within the past 6 months
* Prior major surgery or trauma within 28 days prior to first dose of study drug, and/or not recovered from effects of that surgery, and/or presences of an non-healing wound, fracture or ulcer, or patients that may require surgery during the course of treatment
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions or involvement of large pulmonary vessels by tumor
* Hemoptysis within 6 weeks of the first dose of study drug
* Clinically significant gastrointestinal abnormalities that may increase the risk of GI bleeding
* Expansion Cohort Only: Currently active second malignancy other than non-melanoma skin cancers
* Presence of uncontrolled infection
* Liver disease such as chronic cirrhosis, active hepatitis or chronic persistent hepatitis
* Uncontrolled diabetes
* Pregnant or breastfeeding
* Chronic treatment with systemic corticosteroids or other immunosuppressive agent
* Treatment with strong CYP3A4 inhibitors
* Treatment with strong CYP3A4 inducers
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Prolongation of corrected QT interval > 480msecs
* History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of stomach or small bowel that could interfere with absorption, distribution, metabolism, or excretion of study drugs
* Any ongoing toxicity from prior anti-cancer therapy that is greater than grade 1 and/or that is progressing in severity.
* Any serious and/or pre-existing medical, psychiatric, or other condition that could interfere with subject safety, obtaining informed consent or compliance with study procedures
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pomerantz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellmunt J, Lalani AA, Jacobus S, Wankowicz SA, Polacek L, Takeda DY, Harshman LC, Wagle N, Moreno I, Lundgren K, Bosse D, Van Allen EM, Choueiri TK, Rosenberg JE. Everolimus and pazopanib (E/P) benefit genomically selected patients with metastatic urothelial carcinoma. Br J Cancer. 2018 Sep;119(6):707-712. doi: 10.1038/s41416-018-0261-0. Epub 2018 Sep 17. PMID 30220708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between January 2011 and July 2016 including dose finding 1/1/2011-9/23/2011 and expansion 3/9/2015-7/25/2016.
Period: Overall Study
Arm/Group | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg | All Phase I Dose Expansion Participants
Started | 3 | 6 | 14
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed'.) | 0 | 0 | 0
Not Completed | 3 | 6 | 14
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Disease Progression | 1 | 3 | 12

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg | All Phase I Dose Expansion Participants | Total
Number analyzed (Participants) | 3 | 6 | 14 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [50 to 77] | 58 [50 to 61] | 69 [66 to 72] | 66 [59 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 2 | 6
  Male | 3 | 2 | 12 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1 | 2
  White | 3 | 5 | 13 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 14 | 23
Tumor type [Count of Participants; unit: Participants]
  Adrenal cortex | 0 | 1 | 0 | 1
  Bladder | 3 | 2 | 14 | 19
  Lung | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) [Phase I Dose Finding]
Description: The MTD of Pazopanib in combination with Everolimus 5 mg PO QD was determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached.
Time Frame: Participants were assessed for adverse events on days 1 and 15 for cycles 1-2 and every cycle thereafter; The observation period for MTD evaluation was the first 28 days of treatment.
Population: All phase I dose finding participants who received at least one dose of the study drug were evaluable for MTD.
Measure: Number; unit: mg
Groups:
- All Phase I Dose Finding Participants: All phase I dose finding participants received Everolimus 5mg and Pazopanib according to the established dose escalation schedule.
Arm/Group | All Phase I Dose Finding Participants
Number analyzed (Participants) | 9
mg | 400

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I Dose Finding]
Description: A DLT was defined as an adverse event (a) with treatment attribution of possible, probable, or definite, and (b) occurs during cycle 1, and (c) meets any of the following criteria: Grade 3 or 4 non-hematologic toxicity excluding: nausea/vomiting controlled with antiemetics, Grade 3 hypertension that resolves to ≤150/90 within 7 days with supportive care, and Grade 3 asymptomatic, clinically insignificant laboratory abnormalities (LDH, alkaline phosphatase due to bone metastases, and asymptomatic hypophosphatemia). Hematologic toxicity: Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with bleeding, Grade 4 neutropenia which persists for >7 days, Grade 4 neutropenia associated with fever >38.5C; Hematologic toxicity excluded lymphopenia or anemia of any grade. Missing more than 5 days of planned doses for drug-related intolerable grade 2 toxicity;Toxicity related to therapy severe enough to require a dose-reduction.
Time Frame: Participants were assessed for adverse events on days 1 and 15 for cycles 1-2 and every cycle thereafter; The observation period for DLT evaluation was the first 28 days of treatment.
Population: All phase I dose finding participants who received at least one dose of the study drug were evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg
Number analyzed (Participants) | 3 | 6
Participants | 2 | 0

3. Primary Outcome: Objective Response Rate [Expansion]
Description: The objective response rate (ORR) was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: TDisease was evaluated radiologically at baseline and every 8 weeks on treatment; Treatment duration was up to 6 cycles in the Dose Level 0 cohort, 14 cycles in the Dose Level -1 cohort and 10 cycles in the expansion cohort (1 cycle=28 days).
Population: The analysis population is comprised of all enrolled Phase 1 expansion participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Phase I Dose Expansion Participants
Number analyzed (Participants) | 14
percentage of participants | 21.4 [4.7 to 50.8]

4. Secondary Outcome: Grade 4 Treatment-Related Toxicity Rate [Dose Finding]
Description: Grade 4 treatment-related toxicity rate is the percentage of participants experiencing at least one treatment-related grade 4 adverse event (AE) with treatment attribution of possibly, probably or definite based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) as reported on case report forms.
Time Frame: Participants were assessed for adverse events on days 1 and 15 for cycles 1-2 and every cycle thereafter; Treatment duration was up to 6 cycles in the Dose Level 0 cohort and 14 cycles in the Dose Level -1 cohort (1 cycle=28 days).
Population: All phase I dose finding participants who received at least one dose of the study drug were evaluable for toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Level 0: Everolimus 5mg + Pazopanib 600 mg [Dose Finding]: Everolimus 5mg + Pazopanib 600 mg once daily for 28 days each cycle Participants were treated until disease progression, unacceptable toxicity or patient withdrawal.
- Dose Level -1: Everolimus 5mg + Pazopanib 400 mg [Dose Finding: Everolimus 5mg + Pazopanib 400 mg once daily for 28 days each cycle Participants were treated until disease progression, unacceptable toxicity or patient withdrawal.
Arm/Group | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg [Dose Finding] | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg [Dose Finding
Number analyzed (Participants) | 3 | 6
percentage of participants | 33.3 [0.9 to 90.6] | 0.0 [0.0 to 45.9]

5. Secondary Outcome: Median Progression-Free Survival [Expansion]
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Participants alive without PD are censored at date of last disease assessment. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum longest diameter (LD), taking as reference the smallest sum on study with at least 5 mm absolute increase or the appearance of one or more new lesions. For non-target lesions, PD is appearance of one or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; PFS follow-up was up to 9.2 months in the expansion cohort.
Population: The analysis population is comprised of all enrolled Phase 1 expansion participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Phase I Dose Expansion Participants
Number analyzed (Participants) | 14
months | 2.9 [0.9 to 3.6]

6. Secondary Outcome: Mean Duration of Response [Expansion]
Description: Duration of response was calculated as the time from achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment until disease progression. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. For target lesions: PD is at least a 20% increase in sum longest diameter (LD), taking as reference the smallest sum on study with at least 5 mm absolute increase or the appearance of one or more new lesions. For non-target lesions, PD is appearance of one or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 5
Population: The duration of response is only estimated in the phase 1 expansion participants who achieved objective response on treatment.
Measure: Mean (Full Range); unit: months
Arm/Group | All Phase I Dose Expansion Participants
Number analyzed (Participants) | 14
months | 4.9 [1.7 to 7.4]

7. Secondary Outcome: Grade 4 Treatment-Related Toxicity Rate [Expansion]
Description: as for outcome 4
Time Frame: Participants were assessed for adverse events on days 1 and 15 for cycles 1-2 and every cycle thereafter; Treatment duration was up to 10 cycles in the expansion cohort (1 cycle=28 days).
Population: All phase I expansion participants who received at least one dose of the study drug were evaluable for toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Phase I Dose Expansion Participants
Number analyzed (Participants) | 14
percentage of participants | 7.1 [0.2 to 33.9]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events on days 1 and 15 for cycles 1-2 and every cycle thereafter; Treatment duration was up to 13 cycles in this study cohort (1 cycle=28 days).
Description: Maximum grade toxicity by type was first calculated. Serious adverse events were defined as events with treatment attribution of possibly, probably, or definitely related and grade 3 or higher per CTCAE v4.0. Other adverse events were defined as grade 1-2 events with treatment attribution of possibly, probably, or definitely related and grades 1-5 with unrelated attribution CTCAE v4.0.
Groups:
- Dose Level -1: Everolimus 5mg + Pazopanib 400 mg; All Phase I Dose Expansion Participants: All phase I dose expansion participants received Everolimus 5mg and Pazopanib at the maximum tolerated dose established in the dose finding part of the study.
Arm/Group | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg | All Phase I Dose Expansion Participants
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/6 | 9/14
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/6 | 13/14
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg (N=3) | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg (N=6) | All Phase I Dose Expansion Participants (N=14)
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2
General disorders and administration site conditions (other) (General disorders) | 1 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0: Everolimus 5mg + Pazopanib 600 mg (N=3) | Dose Level -1: Everolimus 5mg + Pazopanib 400 mg (N=6) | All Phase I Dose Expansion Participants (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 3 | 4
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 6
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Cardiac disorder other (Cardiac disorders) | 0 | 0 | 1
Cholesterol high (Investigations) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 7
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Edema limbs (General disorders) | 0 | 1 | 3
Edema trunk (General disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 5 | 6
GGT increased (Investigations) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Fever (General disorders) | 1 | 2 | 0
General disorders and administration site conditions (other) (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2 | 4
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1
Injury, poisoning and procedural complications (other) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 1
Metabolism and nutrition disorders (other) (Metabolism and nutrition disorders) | 0 | 0 | 1
Mucosal infection (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 3 | 3
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 2
Nervous system disorders (other) (Nervous system disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Phantom pain (Nervous system disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 4 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Serum amylase increased (Investigations) | 0 | 2 | 3
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1
Weight loss (Investigations) | 1 | 2 | 4
White blood cell decreased (Investigations) | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
The phase 1 expansion cohort was terminated early due to weak accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT01184326/Prot_SAP_000.pdf